CLINICAL TRIAL: NCT04759482
Title: Validation of an Innovative Algorithm for Screening Sleep Apnea Syndrome From an Electrocardiographic Recording During Sleep
Brief Title: Validation of a New Algorithm for Screening Sleep Apnea Syndrome From Electrocardiogram
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI046
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Sleep Apnea
Keywords: sleep; electrocardiogram; screening; apnea; polysomnography; algorithm
MeSH Terms: conditions — Sleep Apnea Syndromes; Apnea | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with sleep apnea: We selected 150 patients recorded by polysomnography between january 2019 and june 2020 in the Center for Sleep Medecine and Research in Nancy.
  Interventions: Diagnostic Test: polysomnography

INTERVENTIONS:
Diagnostic Test: polysomnography — Polysomnography consisted in recording sleep parameters during one night, using a non-invasive multi-channels device, including respiratory sensors, electrocardiogram and electroencephalogram

SUMMARY:
Sleep apnea syndrome is a prevalent disease, recognized as an independant risk factor for cardiovascular diseases The gold standard for the diagnosis of sleep apnea is the polysomnography. But polysomnography is time-consuming and very expensive. We developed an algorithm for screening sleep apnea from electrocardiographic signal. This would lead to the simplification of screening sleep apnea by using a two-channels recording device and computerizing the scoring of respiratory events. The validation of the algorithm will consist in comparing the number of apnea and hypopnea per hour of sleep (AHI) detected by the algorithm from the electrocardiographic signal recorded during a standard polysomnography in the Center for Sleep Medicine and Research in Nancy, with the AHI resulted from the standard interpretation of the same polysomnography by experts in sleep scoring (gold standard).

ELIGIBILITY:
Inclusion Criteria:

* all patients with a polysomnography recorded in the Center for Sleep Medecine and Research (CSMR) in Nancy from january 2019 and june 2020
* results of standard interpretation of polysomnography giving a number of hypopnea and apnea per hour of sleep (AHI) superior to 5

Exclusion Criteria:

* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient refered to the CSMR, for which sleep apnea are supected
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Concordance of the number of sleep hypopnea and apnea between an algorithm computerizing the electrocardiographic signal and the standard interpretation of the polysomnography by an expert in sleep scoring (gold standard) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: El Mehdi Siaghy, Study Chair — Research and Innovation Department

IPD SHARING:
Plan to Share IPD: Undecided